CLINICAL TRIAL: NCT03031821
Title: A Randomized Phase 3 Trial of Metformin in Patients Initiating Androgen Deprivation Therapy as Prevention and Intervention of Metabolic Syndrome: The Prime Study
Brief Title: Metformin in Patients Initiating ADT as Prevention and Intervention of Metabolic Syndrome
Acronym: PRIME
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Manufacturer discontinued the production of study drugs.
Sponsor: Canadian Urologic Oncology Group (Other)
Collaborators: Prostate Cancer Canada (Other); British Columbia Cancer Agency (Other); BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRIME
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Metabolic Syndrome
Keywords: Prostate Cancer; ADT; Metabolic Syndrome; Androgen Deprivation Therapy; Phase III; Phase 3; Randomized
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin 850 mg PO OD X 30 days, then 850mg PO BID for a total of 18 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo Oral Tablet
  1 tablet (850mg) PO OD X 30 days, then 850mg PO BID for a total of 18 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin — Metformin Duration: 18 months 850 mg PO OD x 30 days then 850 mg PO BID for duration
  Arms: Metformin
Drug: Placebo Oral Tablet — Placebo Oral Tablet Duration 18 months
  1 tablet (850 mg) PO OD x 30 days then 1 tablet PO BID for duration
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a multi-centre, double-blind, randomized phase III trial comparing metformin to placebo in patients with advanced prostate cancer starting (or have recently started) androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
The primary objective of this study will determine if there are differences between arms with respect to the proportion of participants who meet the diagnostic criteria for metabolic syndrome after 18 months of study treatment.

The investigators will also compare arms with regards to severity of individual metabolic syndrome components following 18 months of study treatment. Other objectives are outlined below, and will include quality of life assessments, metabolic and anthropomorphic measurements at additional time points and correlative laboratory studies.

It is estimated that one in seven Canadian men will be diagnosed with prostate cancer in their lifetime. In 2015, approximately 23,600 Canadian men were estimated to be diagnosed with prostate cancer and 4,000 died of this disease.

Androgen deprivation therapy (ADT) is a standard first-line treatment for men with incurable prostate cancer and has long been known to improve overall survival.

Although the effectiveness of ADT is well established in participants with advanced prostate cancer, it is associated with important adverse effects as outlined below. The development of metabolic syndrome in particular is clinically important as it is associated with worsened quality of life and increased all-cause morbidity and mortality.

As ADT is now employed, alone or in combination with other therapies, in virtually all men with advanced prostate cancer for increasingly long periods of time (median survival of men presenting with newly diagnosed metastatic disease from recent clinical trials is at least 3 years, during which they are typically on continuous hormonal therapy), the burden of ADT toxicity among men with prostate cancer is significant and increasing.

The investigators hypothesize that the addition of metformin to a program of ADT will reduce the proportion of participants with metabolic syndrome at 18 months after initiation of ADT and will reduce the severity of individual components of metabolic syndrome in men with advanced prostate cancer. To test this hypothesis, this is a randomized, double-blinded, placebo-controlled phase 3 clinical trial of metformin in patients undergoing ADT treatment.

ELIGIBILITY:
Inclusion Criteria

Participants must fulfill all the following criteria to be eligible for admission to the study:

1. Pathologically confirmed adenocarcinoma of the prostate
2. Eligible for initiating androgen deprivation therapy with either:

   1. (Neo-)Adjuvant therapy for localized prostate cancer that is planned continuously for at least 9 months; or
   2. Metastatic disease: or
   3. Biochemical recurrence of prostate cancer as defined as EITHER:

      * A rising PSA after prior curative intent surgical therapy (e.g., prostatectomy with or without adjuvant/ salvage radiotherapy). Since an absolute consensus for this value has not been established, if a rising PSA has been documented by at least two PSA values at least 2 weeks apart, the criteria for biochemical recurrence are deemed to have been met. Or,
      * PSA ≥ 2ng/mL above their nadir if previously treated with definitive radiotherapy
3. Serum testosterone > 5nmol/L (except for participants who have already started androgen deprivation therapy (within no more than 45 days of commencing study treatment)).
4. The choice of androgen deprivation therapy is at the investigators discretion but must include at minimum the use of luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy. The addition of other hormonal agents (e.g., non-steroidal antiandrogens, abiraterone, enzalutamide, apalutamide) is allowed.
5. The androgen deprivation therapy undertaken can be intermittent or continuous, but the treatment intent must be declared prior to randomization.
6. Participant is able (e.g., sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French. The baseline assessment must be completed within required timelines, prior to registration/randomization. Inability (lack of comprehension in English or French, or other equivalent reason such as cognitive issues or lack of competency) to complete the questionnaires will not make the participant ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the participant ineligible.
7. Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrolment in the trial to document their willingness to participate.
8. Participant must be accessible for treatment and follow up. Participants registered on this trial must be treated and followed at the participating centre. Investigators must assure themselves that the participants registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
9. Protocol treatment is to begin within 7 working days of participant randomization.

Exclusion Criteria

Participants who fulfill any of the following criteria are not eligible for admission to the study:

1. Prior androgen deprivation therapy within 12 months of enrolment (except for participants who have started androgen deprivation therapy within 45 days of commencing study treatment)

   * Prior androgen deprivation therapy associated with definitive treatment is permitted, if it has been completed at least 12 months prior to enrolment (e.g., last injection or tablet taken 12 months prior to study enrolment)
2. Participant that meet ≥ 1 of the Canadian Diabetes Association criteria for the diagnosis of diabetes within 28 days of enrolment:

   * Fasting plasma glucose of ≥ 7mmol/L; or
   * HbA1C ≥ 6.5%.
3. Participant currently taking metformin (or other diabetic medications) or who have taken metformin (or other diabetic medications) within 28 days of enrolment.
4. History of lactic acidosis or conditions that predispose to lactic acidosis:

   * Impaired Renal Function (eGFR <45mL/ minute/ 1.73 m^2); or
   * Liver disease, including alcoholic liver disease, as demonstrated by any of the following parameters:

     1. AST > 1.8 x the upper limit of normal
     2. ALT > 1.8 x the upper limit of normal
     3. Alkaline Phosphatase >2x the upper limit of normal
     4. Serum total bilirubin > 1.5x the upper limit of normal (except for participant with Gilbert's Disease who are eligible despite elevated serum bilirubin levels).
   * Alcohol abuse (habitual intake of ≥ 3 alcoholic beverages per day) sufficient to cause hepatic toxicity; or
   * Severe infection; or
   * Congestive heart failure (defined as New York Heart Association Class III or IV functional status).
5. Participant with a history of other invasive malignancies, except adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who meet the diagnostic criteria for metabolic syndrome after 18 months of study treatment | 18 months
  A diagnosis of metabolic syndrome will be made according to the harmonized definition of the metabolic syndrome as defined in the joint statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and the International Association for the Study of Obesity. A patient will be classified as having metabolic syndrome if he possesses ≥3 of the aforementioned criteria: Increased waist circumference, elevated triglycerides, reduced high-density lipoprotein cholesterol, elevated blood pressure, and elevated fasting blood glucose.
  The prevalence of metabolic syndrome at 18 months post randomization will be calculated and compared between treatment arms using the two-sample t-test.

SECONDARY OUTCOMES:
Proportion of participants who meet the diagnostic criteria for metabolic syndrome after 9 months of study treatment | 9 months
  A diagnosis of metabolic syndrome will be made according to the harmonized definition of the metabolic syndrome as defined in the joint statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and the International Association for the Study of Obesity. A patient will be classified as having metabolic syndrome if he possesses ≥3 of the aforementioned criteria: Increased waist circumference, elevated triglycerides, reduced high-density lipoprotein cholesterol, elevated blood pressure, and elevated fasting blood glucose.
  The prevalence of metabolic syndrome at 9 months post randomization will be calculated and compared between treatment arms using the two-sample t-test.
Proportion of participants who meet the diagnostic criteria for metabolic syndrome after 12 months of study treatment | 12 months
  A diagnosis of metabolic syndrome will be made according to the harmonized definition of the metabolic syndrome as defined in the joint statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and the International Association for the Study of Obesity. A patient will be classified as having metabolic syndrome if he possesses ≥3 of the aforementioned criteria: Increased waist circumference, elevated triglycerides, reduced high-density lipoprotein cholesterol, elevated blood pressure, and elevated fasting blood glucose.
  The prevalence of metabolic syndrome at 12 months post randomization will be calculated and compared between treatment arms using the two-sample t-test.
Proportion of participants who meet the diagnostic criteria for metabolic syndrome after 24 months of study treatment | 24 months
  A diagnosis of metabolic syndrome will be made according to the harmonized definition of the metabolic syndrome as defined in the joint statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and the International Association for the Study of Obesity. A patient will be classified as having metabolic syndrome if he possesses ≥3 of the aforementioned criteria: Increased waist circumference, elevated triglycerides, reduced high-density lipoprotein cholesterol, elevated blood pressure, and elevated fasting blood glucose.
  The prevalence of metabolic syndrome at 24 months post randomization will be calculated and compared between treatment arms using the two-sample t-test.
Proportion of participants who meet the criteria of reduced high-density lipoprotein cholesterol assessed at 18 months of follow-up. | 18 months
  Reduced High-Density Lipoprotein Cholesterol defined as: < 1.0 mmol/L; or drug treatment for reduced HDL cholesterol*
  *Patient taking fibrates (Bezafibrate, Ciprofibrate, Clofibrate, Gemfibrozil, or Fenofibrate) or nicotinic acid can be presumed to have high TG and reduced HDL-cholesterol levels; Patients taking high dose omega-3 fatty acids can be presumed to have high TG levels
Proportion of participants who meet the criteria of elevated triglycerides assessed at 18 months of follow-up. | 18 months
  Elevated Triglycerides defined as: ≥1.7 mmol/L; or drug treatment for elevated triglycerides*
  *Patient taking fibrates (Bezafibrate, Ciprofibrate, Clofibrate, Gemfibrozil, or Fenofibrate) or nicotinic acid can be presumed to have high TG and reduced HDL-cholesterol levels; Patients taking high dose omega-3 fatty acids can be presumed to have high TG levels
Proportion of participants who meet the criteria of elevated blood pressure assessed at 18 months of follow-up. | 18 months
  Elevated Blood Pressure defined as:
  Systolic Blood Pressure of ≥ 130 mm of Hg; or Diastolic Blood Pressure of ≥ 85 mm of Hg; or drug treatment for elevated blood pressure
  Blood pressures will be taken with patients sitting for 5 minutes in a quiet environment prior to measurement and two measurements taken (with a minimum of 5 minutes between each blood pressure measurement), with the mean recorded for this study.
Proportion of participants who meet the criteria of elevated fasting blood glucose levels assessed at 18 months of follow-up. | 18 months
  Elevated Fasting Blood Glucose defined as:
  HbA1c ≥ 6.5%; or Fasting plasma glucose ≥ 7.0 mmol/L; or drug treatment for elevated blood glucose
Proportion of participants who meet the criteria of increased waist circumference assessed at 18 months of follow-up. | 18 months
  Increased Waist Circumference defined as:
  Males (population and country specific) A) Canadians ≥102cm B) Chinese ≥ 85cm C) Japanese ≥ 85 cm D) Other Asians ≥ 90 cm E) Middle Eastern & Mediterranean ≥ 94cm F) Sub-Saharan African ≥ 94 cm G) Central & South American ≥ 90cm H) Europid ≥ 94 cm
  Measurement of waist circumference will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Health-related Quality of Life assessed at 18 months of follow-up. | 18 months
  Patients will undergo quality of life measurements by the EORTC QLQ-C30 core questionnaire (63) and prostate-specific module. The instruments are well validated and widely used in the population of interest. The questionnaire items are transformed for 5 functional domains, global QOL, and specific symptom scales/items relevant to the study intervention.
  The statistical analysis plan will use the standard CCTG QOL approach (Osoba et al., 1998), and will focus on change of mean scores from baseline over time by treatment allocation group. Depending on the amount of missing data, generalized linear equation modeling of mean scores may be required. The analysis will also consider the proportion of patients improved, stable or deteriorated at 18 months compared to baseline using a cut-point minimal clinical difference of 10 points on all scales. A sensitivity analysis will be executed using a cut-point of 7 points.
Treatment-related toxicity | 18 months
  Treatment related toxicity (NCI CTCAE 4.0)
  All men will be evaluated for toxicity from the time of their first oral dose of study medication. Toxicities will be graded using the current CTCAE version 4.0. The incidence of toxicities by arm will be summarized by type of adverse effect. A Fisher's Exact Test will be used to compare toxicities between the two arms.

OTHER OUTCOMES:
Serum insulin levels assessed at 18 months of follow-up. | 18 months
  Fasting insulin level
  Test for significance: Two sample independent t-test.
Insulin resistance assessed at 18 months of follow-up. | 18 months
  The homoeostasis model assessment insulin resistance (HOMA-IR) (67, 68) and the Quantitative Insulin Sensitivity Check Index (QUICKI) (69), indirect measures of insulin resistance, will be the primary means of classifying insulin resistance status for this study.
  HOMA-IR = Fasting Insulin (μU/ml) * Fasting glucose (mmol/L) 22.5
  QUICKI = 1/[log fasting insulin (mU/L) + log fasting glucose (mg/dl)]
Time to re-initiation of androgen deprivation therapy (in the subset of patients receiving intermittent therapy) | 18 months
  The median duration of time off-treatment (i.e. ADT) in days will be compared between study arms using the student t-test.
Duration of time off-treatment in days | 18 months
  The median duration of time off-treatment (i.e. ADT) in days will be compared between study arms (in the subset of patients on intermittent ADT) using the student t-test.
Testosterone levels assessed at 18 months of follow-up. | 18 months
  Testosterone to be measured as per standard of care (usually every 3 months during initiation of ADT and initial off-ADT period).
Body mass assessed at 18 months of follow-up. | 18 months
  Measurement weight will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Abdominal girth assessed at 18 months of follow-up. | 18 months
  Measurement of abdominal girth will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Mean BMI assessed at 12 months of follow-up. | 12 months
  Measurement of height and weight will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Mean BMI assessed at 24 months of follow-up. | 24 months
  Measurement of height and weight will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Mean BMI assessed at 36 months of follow-up. | 36 months
  Measurement of height and weight will be performed by a dedicated research nurse for this study that is blinded to the patient's treatment allocation.
Exercise behavior and sedentary behavior assessed at 12 months of follow-up. | 12 months
  Exercise/sedentary questionnaire will be administered at 12 months of follow-up.
  Analyses of covariance (ANCOVA) to explore the effects of the intervention on moderate exercise minutes, vigorous exercise minutes, combined moderate and vigorous exercise minutes, and sedentary behavior hours will be conducted. Chi-square analyses to examine the effects of the intervention on meeting the exercise guidelines will be done.
Exercise behavior and sedentary behavior assessed at 24 months of follow-up. | 24 months
  Exercise/sedentary questionnaire will be administered at 24 months of follow-up.
  Analyses of covariance (ANCOVA) to explore the effects of the intervention on moderate exercise minutes, vigorous exercise minutes, combined moderate and vigorous exercise minutes, and sedentary behavior hours will be conducted. Chi-square analyses to examine the effects of the intervention on meeting the exercise guidelines will be done.
Exercise behavior and sedentary behavior assessed at 36 months of follow-up. | 36 months
  Exercise/sedentary questionnaire will be administered at 36 months of follow-up.
  Analyses of covariance (ANCOVA) to explore the effects of the intervention on moderate exercise minutes, vigorous exercise minutes, combined moderate and vigorous exercise minutes, and sedentary behavior hours will be conducted. Chi-square analyses to examine the effects of the intervention on meeting the exercise guidelines will be done.
Cardiovascular mortality | Through study completion, an average of 3 years
  For cardiovascular morality, the survival period will be defined as the date of randomization to the date of death due to cardiovascular disease or the date of censoring. All deaths that occur amongst study participants will be reviewed by the study's data safety and monitoring committee (who will be blinded to the treatment allocation of the patient in question). Deaths will be classified into 3 categories: 1) Prostate Cancer 2) Cardiovascular Disease 3) Other. Cardiovascular deaths will include cases in which cardiovascular disease, coronary artery disease, or stroke are identified as one of the causes of death, not just the underlying cause of death.
Biochemical progression-free survival | 36 months
  For bPFS, the survival period will be defined as the date of randomization to the date of biochemical progression or the date of censoring. For the purposes of this study, biochemical progression will be defined as a rise in serum PSA above their pre-randomization level (or 10ng/mL for patients who had a baseline PSA >10ng/mL) or the initiation of cancer treatment (i.e. second course of hormonal therapy, systemic therapy, etc.).
Castration resistant disease-free survival | 36 months
  For RFS-CR, the survival period will be defined as the date of randomization to the date of confirmed biochemical castration resistance or the date of censoring. For the purposes of this study, castration resistance will be defined as a continuous rise in serum PSA despite castrate levels of serum testosterone (achieved via total androgen blockade).
Distant metastasis disease-free survival | 36 months
  For RFS-DM, the survival period will be defined as the date of randomization to the date of confirmation of distant metastases or the date of censoring. Any of the following constitute a confirmation of distant metastases: imaging evidence of de novo bone metastases (X-rays, bone scan, CT, MRI, or PET scan), pathological fracture secondary to a bone metastases, imaging evidence of lymph node metastases (CT, MRI or Ultrasound Scans).
Prostate cancer specific survival | Through study completion, an average of 3 years
  For PCSS, the survival period will be defined as the date of randomization to the date of death due to prostate cancer or the date of censoring. All deaths that occur amongst study participants will be reviewed by the study's data safety and monitoring committee (who will be blinded to the study arm allocation of the patient in question). Any death that is determined to be attributable to a participant's prostate cancer will be deemed a death due to prostate cancer.
Overall survival | Through study completion, an average of 3 years
  For OS, the survival period will be defined as the date of randomization to the date of death due to any cause or the date of censoring. All deaths that occur amongst study participants will be reviewed by the study's data safety and monitoring committee (who will be blinded to the treatment allocation of the patient in question). Deaths will be classified into 3 categories: 1) Prostate Cancer 2) Cardiovascular Disease 3) Other.

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Eigl, MD, Study Chair — British Columbia Cancer Agency; Nawaid Usmani, MD, Study Chair — University of Alberta
Locations (16):
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnepeg, Manitoba
  - Horizon Health Network, Saint John, New Brunswick
  - Central Newfoundland Regional Health Centre, Grand Falls-Windsor, Newfoundland and Labrador
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Northeast Cancer Centre, Greater Sudbury, Ontario
  - Sunnybrook Research Institue, Toronto, Ontario
  - Princess Margaret Cancer Centre (Princess Margaret Hospital), Toronto, Ontario
  - CHU de Quebec - Universite Laval, Laval, Quebec
  - Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Center-Cedar Cancer Center, Montreal, Quebec
  - Ciusss-Chus, Sherbrooke, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Mauricie-Centre-du-Québec / Centre hospitalier régional, Trois-Rivières, Quebec

REFERENCES:
- [Background] Canadian Cancer Society. Canadian Cancer Statistics 2015: Canadian Cancer Society; 2015 [Available from: http://www.cancer.ca/].
- [Background] Crook JM, O'Callaghan CJ, Duncan G, Dearnaley DP, Higano CS, Horwitz EM, Frymire E, Malone S, Chin J, Nabid A, Warde P, Corbett T, Angyalfi S, Goldenberg SL, Gospodarowicz MK, Saad F, Logue JP, Hall E, Schellhammer PF, Ding K, Klotz L. Intermittent androgen suppression for rising PSA level after radiotherapy. N Engl J Med. 2012 Sep 6;367(10):895-903. doi: 10.1056/NEJMoa1201546. PMID 22931259
- [Background] Hussain M, Tangen CM, Berry DL, Higano CS, Crawford ED, Liu G, Wilding G, Prescott S, Kanaga Sundaram S, Small EJ, Dawson NA, Donnelly BJ, Venner PM, Vaishampayan UN, Schellhammer PF, Quinn DI, Raghavan D, Ely B, Moinpour CM, Vogelzang NJ, Thompson IM Jr. Intermittent versus continuous androgen deprivation in prostate cancer. N Engl J Med. 2013 Apr 4;368(14):1314-25. doi: 10.1056/NEJMoa1212299. PMID 23550669
- [Background] Lakka HM, Laaksonen DE, Lakka TA, Niskanen LK, Kumpusalo E, Tuomilehto J, Salonen JT. The metabolic syndrome and total and cardiovascular disease mortality in middle-aged men. JAMA. 2002 Dec 4;288(21):2709-16. doi: 10.1001/jama.288.21.2709. PMID 12460094
- [Background] Malik S, Wong ND, Franklin SS, Kamath TV, L'Italien GJ, Pio JR, Williams GR. Impact of the metabolic syndrome on mortality from coronary heart disease, cardiovascular disease, and all causes in United States adults. Circulation. 2004 Sep 7;110(10):1245-50. doi: 10.1161/01.CIR.0000140677.20606.0E. Epub 2004 Aug 23. PMID 15326067
- [Background] Mottillo S, Filion KB, Genest J, Joseph L, Pilote L, Poirier P, Rinfret S, Schiffrin EL, Eisenberg MJ. The metabolic syndrome and cardiovascular risk a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Sep 28;56(14):1113-32. doi: 10.1016/j.jacc.2010.05.034. PMID 20863953
- [Background] Solymoss BC, Bourassa MG, Campeau L, Sniderman A, Marcil M, Lesperance J, Levesque S, Varga S. Effect of increasing metabolic syndrome score on atherosclerotic risk profile and coronary artery disease angiographic severity. Am J Cardiol. 2004 Jan 15;93(2):159-64. doi: 10.1016/j.amjcard.2003.09.032. PMID 14715340
- [Background] Miettola J, Niskanen LK, Viinamaki H, Sintonen H, Kumpusalo E. Metabolic syndrome is associated with impaired health-related quality of life: Lapinlahti 2005 study. Qual Life Res. 2008 Oct;17(8):1055-62. doi: 10.1007/s11136-008-9386-6. Epub 2008 Aug 31. PMID 18759109
- [Background] Park SS, Yoon YS, Oh SW. Health-related quality of life in metabolic syndrome: The Korea National Health and Nutrition Examination Survey 2005. Diabetes Res Clin Pract. 2011 Mar;91(3):381-8. doi: 10.1016/j.diabres.2010.11.010. Epub 2010 Dec 4. PMID 21134699
- [Background] Ford ES, Li C. Metabolic syndrome and health-related quality of life among U.S. adults. Ann Epidemiol. 2008 Mar;18(3):165-71. doi: 10.1016/j.annepidem.2007.10.009. PMID 18280918
- [Background] Nguyen PL, Alibhai SM, Basaria S, D'Amico AV, Kantoff PW, Keating NL, Penson DF, Rosario DJ, Tombal B, Smith MR. Adverse effects of androgen deprivation therapy and strategies to mitigate them. Eur Urol. 2015 May;67(5):825-36. doi: 10.1016/j.eururo.2014.07.010. Epub 2014 Aug 2. PMID 25097095
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Mohler JL, Armstrong AJ, Bahnson RR, D'Amico AV, Davis BJ, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Kane CJ, Kawachi MH, Kuettel M, Lee RJ, Meeks JJ, Penson DF, Plimack ER, Pow-Sang JM, Raben D, Richey S, Roach M 3rd, Rosenfeld S, Schaeffer E, Skolarus TA, Small EJ, Sonpavde G, Srinivas S, Strope SA, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 1.2016. J Natl Compr Canc Netw. 2016 Jan;14(1):19-30. doi: 10.6004/jnccn.2016.0004. PMID 26733552
- [Background] Kylin E. Studien ueber das Hypertonie-Hyperglykaemie-Hyperurikaemiesydrom. Zentralblatt fuer Innere Medizin. 1923;44:105-27.
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Kaplan NM. The deadly quartet and the insulin resistance syndrome: an historical overview. Hypertens Res. 1996 Jun;19 Suppl 1:S9-11. doi: 10.1291/hypres.19.supplementi_s9. PMID 9240756
- [Background] Haffner SM, Valdez RA, Hazuda HP, Mitchell BD, Morales PA, Stern MP. Prospective analysis of the insulin-resistance syndrome (syndrome X). Diabetes. 1992 Jun;41(6):715-22. doi: 10.2337/diab.41.6.715. PMID 1587398
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Tsai HK, D'Amico AV, Sadetsky N, Chen MH, Carroll PR. Androgen deprivation therapy for localized prostate cancer and the risk of cardiovascular mortality. J Natl Cancer Inst. 2007 Oct 17;99(20):1516-24. doi: 10.1093/jnci/djm168. Epub 2007 Oct 9. PMID 17925537
- [Background] Braga-Basaria M, Dobs AS, Muller DC, Carducci MA, John M, Egan J, Basaria S. Metabolic syndrome in men with prostate cancer undergoing long-term androgen-deprivation therapy. J Clin Oncol. 2006 Aug 20;24(24):3979-83. doi: 10.1200/JCO.2006.05.9741. PMID 16921050
- [Background] Cleffi S, Neto AS, Reis LO, Maia P, Fonseca F, Wroclawski ML, Neves M, Pompeo AC, Del Giglio A, Faria EF, Tobias-Machado M. [Androgen deprivation therapy and morbid obesity: do they share cardiovascular risk through metabolic syndrome?]. Actas Urol Esp. 2011 May;35(5):259-65. doi: 10.1016/j.acuro.2011.01.011. Epub 2011 Apr 2. Spanish. PMID 21459486
- [Background] Morote J, Ropero J, Planas J, Celma A, Placer J, Ferrer R, de Torres I. Metabolic syndrome in patients with prostate cancer undergoing androgen suppression. Actas Urol Esp. 2014 Jun;38(5):285-9. doi: 10.1016/j.acuro.2013.09.008. Epub 2013 Dec 20. English, Spanish. PMID 24360772
- [Background] Bosco C, Crawley D, Adolfsson J, Rudman S, Van Hemelrijck M. Quantifying the evidence for the risk of metabolic syndrome and its components following androgen deprivation therapy for prostate cancer: a meta-analysis. PLoS One. 2015 Mar 20;10(3):e0117344. doi: 10.1371/journal.pone.0117344. eCollection 2015. PMID 25794005
- [Background] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238
- [Background] Carmack Taylor CL, Demoor C, Smith MA, Dunn AL, Basen-Engquist K, Nielsen I, Pettaway C, Sellin R, Massey P, Gritz ER. Active for Life After Cancer: a randomized trial examining a lifestyle physical activity program for prostate cancer patients. Psychooncology. 2006 Oct;15(10):847-62. doi: 10.1002/pon.1023. PMID 16447306
- [Background] Basaria S, Muller DC, Carducci MA, Egan J, Dobs AS. Hyperglycemia and insulin resistance in men with prostate carcinoma who receive androgen-deprivation therapy. Cancer. 2006 Feb 1;106(3):581-8. doi: 10.1002/cncr.21642. PMID 16388523
- [Background] Tsai HT, Keating NL, Van Den Eeden SK, Haque R, Cassidy-Bushrow AE, Ulcickas Yood M, Smith MR, Potosky AL. Risk of diabetes among patients receiving primary androgen deprivation therapy for clinically localized prostate cancer. J Urol. 2015 Jun;193(6):1956-62. doi: 10.1016/j.juro.2014.12.027. Epub 2014 Dec 15. PMID 25524243
- [Background] Keating NL, Liu PH, O'Malley AJ, Freedland SJ, Smith MR. Androgen-deprivation therapy and diabetes control among diabetic men with prostate cancer. Eur Urol. 2014 Apr;65(4):816-24. doi: 10.1016/j.eururo.2013.02.023. Epub 2013 Feb 22. PMID 23453420
- [Background] Cox ME, Gleave ME, Zakikhani M, Bell RH, Piura E, Vickers E, Cunningham M, Larsson O, Fazli L, Pollak M. Insulin receptor expression by human prostate cancers. Prostate. 2009 Jan 1;69(1):33-40. doi: 10.1002/pros.20852. PMID 18785179
- [Background] Foretz M, Guigas B, Bertrand L, Pollak M, Viollet B. Metformin: from mechanisms of action to therapies. Cell Metab. 2014 Dec 2;20(6):953-66. doi: 10.1016/j.cmet.2014.09.018. Epub 2014 Oct 30. PMID 25456737
- [Background] Bridges HR, Jones AJ, Pollak MN, Hirst J. Effects of metformin and other biguanides on oxidative phosphorylation in mitochondria. Biochem J. 2014 Sep 15;462(3):475-87. doi: 10.1042/BJ20140620. PMID 25017630
- [Background] Pollak M. Overcoming Drug Development Bottlenecks With Repurposing: Repurposing biguanides to target energy metabolism for cancer treatment. Nat Med. 2014 Jun;20(6):591-3. doi: 10.1038/nm.3596. No abstract available. PMID 24901568
- [Background] Pollak M. Potential applications for biguanides in oncology. J Clin Invest. 2013 Sep;123(9):3693-700. doi: 10.1172/JCI67232. Epub 2013 Sep 3. PMID 23999444
- [Background] Martin-Montalvo A, Mercken EM, Mitchell SJ, Palacios HH, Mote PL, Scheibye-Knudsen M, Gomes AP, Ward TM, Minor RK, Blouin MJ, Schwab M, Pollak M, Zhang Y, Yu Y, Becker KG, Bohr VA, Ingram DK, Sinclair DA, Wolf NS, Spindler SR, Bernier M, de Cabo R. Metformin improves healthspan and lifespan in mice. Nat Commun. 2013;4:2192. doi: 10.1038/ncomms3192. PMID 23900241
- [Background] Pollak MN. Investigating metformin for cancer prevention and treatment: the end of the beginning. Cancer Discov. 2012 Sep;2(9):778-90. doi: 10.1158/2159-8290.CD-12-0263. Epub 2012 Aug 27. PMID 22926251
- [Background] Nobes JP, Langley SE, Klopper T, Russell-Jones D, Laing RW. A prospective, randomized pilot study evaluating the effects of metformin and lifestyle intervention on patients with prostate cancer receiving androgen deprivation therapy. BJU Int. 2012 May;109(10):1495-502. doi: 10.1111/j.1464-410X.2011.10555.x. Epub 2011 Sep 20. PMID 21933330
- [Background] Venkateswaran V, Haddad AQ, Fleshner NE, Fan R, Sugar LM, Nam R, Klotz LH, Pollak M. Association of diet-induced hyperinsulinemia with accelerated growth of prostate cancer (LNCaP) xenografts. J Natl Cancer Inst. 2007 Dec 5;99(23):1793-800. doi: 10.1093/jnci/djm231. Epub 2007 Nov 27. PMID 18042933
- [Background] Joshua AM, Zannella VE, Downes MR, Bowes B, Hersey K, Koritzinsky M, Schwab M, Hofmann U, Evans A, van der Kwast T, Trachtenberg J, Finelli A, Fleshner N, Sweet J, Pollak M. A pilot 'window of opportunity' neoadjuvant study of metformin in localised prostate cancer. Prostate Cancer Prostatic Dis. 2014 Sep;17(3):252-8. doi: 10.1038/pcan.2014.20. Epub 2014 May 27. PMID 24861559
- [Background] Sherifali D, Nerenberg K, Pullenayegum E, Cheng JE, Gerstein HC. The effect of oral antidiabetic agents on A1C levels: a systematic review and meta-analysis. Diabetes Care. 2010 Aug;33(8):1859-64. doi: 10.2337/dc09-1727. Epub 2010 May 18. PMID 20484130
- [Background] Bailey CJ, Turner RC. Metformin. N Engl J Med. 1996 Feb 29;334(9):574-9. doi: 10.1056/NEJM199602293340906. No abstract available. PMID 8569826
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Hong J, Zhang Y, Lai S, Lv A, Su Q, Dong Y, Zhou Z, Tang W, Zhao J, Cui L, Zou D, Wang D, Li H, Liu C, Wu G, Shen J, Zhu D, Wang W, Shen W, Ning G; SPREAD-DIMCAD Investigators. Effects of metformin versus glipizide on cardiovascular outcomes in patients with type 2 diabetes and coronary artery disease. Diabetes Care. 2013 May;36(5):1304-11. doi: 10.2337/dc12-0719. Epub 2012 Dec 10. PMID 23230096
- [Background] United Kingdom Prospective Diabetes Study 24: a 6-year, randomized, controlled trial comparing sulfonylurea, insulin, and metformin therapy in patients with newly diagnosed type 2 diabetes that could not be controlled with diet therapy. United Kingdom Prospective Diabetes Study Group. Ann Intern Med. 1998 Feb 1;128(3):165-75. doi: 10.7326/0003-4819-128-3-199802010-00001. PMID 9454524
- [Background] United Kingdom Prospective Diabetes Study (UKPDS). 13: Relative efficacy of randomly allocated diet, sulphonylurea, insulin, or metformin in patients with newly diagnosed non-insulin dependent diabetes followed for three years. BMJ. 1995 Jan 14;310(6972):83-8. PMID 7833731
- [Background] Hermann LS, Schersten B, Bitzen PO, Kjellstrom T, Lindgarde F, Melander A. Therapeutic comparison of metformin and sulfonylurea, alone and in various combinations. A double-blind controlled study. Diabetes Care. 1994 Oct;17(10):1100-9. doi: 10.2337/diacare.17.10.1100. PMID 7821128
- [Background] Orchard TJ, Temprosa M, Goldberg R, Haffner S, Ratner R, Marcovina S, Fowler S; Diabetes Prevention Program Research Group. The effect of metformin and intensive lifestyle intervention on the metabolic syndrome: the Diabetes Prevention Program randomized trial. Ann Intern Med. 2005 Apr 19;142(8):611-9. doi: 10.7326/0003-4819-142-8-200504190-00009. PMID 15838067
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Ma J, Li H, Giovannucci E, Mucci L, Qiu W, Nguyen PL, Gaziano JM, Pollak M, Stampfer MJ. Prediagnostic body-mass index, plasma C-peptide concentration, and prostate cancer-specific mortality in men with prostate cancer: a long-term survival analysis. Lancet Oncol. 2008 Nov;9(11):1039-47. doi: 10.1016/S1470-2045(08)70235-3. Epub 2008 Oct 3. PMID 18835745
- [Background] Spratt DE, Zhang C, Zumsteg ZS, Pei X, Zhang Z, Zelefsky MJ. Metformin and prostate cancer: reduced development of castration-resistant disease and prostate cancer mortality. Eur Urol. 2013 Apr;63(4):709-16. doi: 10.1016/j.eururo.2012.12.004. Epub 2012 Dec 14. PMID 23287698
- [Background] Margel D, Urbach DR, Lipscombe LL, Bell CM, Kulkarni G, Austin PC, Fleshner N. Metformin use and all-cause and prostate cancer-specific mortality among men with diabetes. J Clin Oncol. 2013 Sep 1;31(25):3069-75. doi: 10.1200/JCO.2012.46.7043. Epub 2013 Aug 5. PMID 23918942
- [Background] Rothermundt C, Hayoz S, Templeton AJ, Winterhalder R, Strebel RT, Bartschi D, Pollak M, Lui L, Endt K, Schiess R, Ruschoff JH, Cathomas R, Gillessen S. Metformin in chemotherapy-naive castration-resistant prostate cancer: a multicenter phase 2 trial (SAKK 08/09). Eur Urol. 2014 Sep;66(3):468-74. doi: 10.1016/j.eururo.2013.12.057. Epub 2014 Jan 4. PMID 24412228
- [Background] Johnson NP. Metformin use in women with polycystic ovary syndrome. Ann Transl Med. 2014 Jun;2(6):56. doi: 10.3978/j.issn.2305-5839.2014.04.15. PMID 25333031
- [Background] Generali JA, Cada DJ. Metformin: prevention and treatment of antipsychotic-induced weight gain. Hosp Pharm. 2013 Oct;48(9):734-77. doi: 10.1310/hpj4809-734. PMID 24421546
- [Background] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2013 Jan;189(1 Suppl):S34-42; discussion S43-4. doi: 10.1016/j.juro.2012.11.017. PMID 23234628
- [Background] Forslund K, Hildebrand F, Nielsen T, Falony G, Le Chatelier E, Sunagawa S, Prifti E, Vieira-Silva S, Gudmundsdottir V, Pedersen HK, Arumugam M, Kristiansen K, Voigt AY, Vestergaard H, Hercog R, Costea PI, Kultima JR, Li J, Jorgensen T, Levenez F, Dore J; MetaHIT consortium; Nielsen HB, Brunak S, Raes J, Hansen T, Wang J, Ehrlich SD, Bork P, Pedersen O. Disentangling type 2 diabetes and metformin treatment signatures in the human gut microbiota. Nature. 2015 Dec 10;528(7581):262-266. doi: 10.1038/nature15766. Epub 2015 Dec 2. PMID 26633628
- [Background] Feig DS, Moses RG. Metformin therapy during pregnancy: good for the goose and good for the gosling too? Diabetes Care. 2011 Oct;34(10):2329-30. doi: 10.2337/dc11-1153. No abstract available. PMID 21949224
- [Background] Brackett CC. Clarifying metformin's role and risks in liver dysfunction. J Am Pharm Assoc (2003). 2010 May-Jun;50(3):407-10. doi: 10.1331/JAPhA.2010.08090. PMID 20452916
- [Background] Lipska KJ, Bailey CJ, Inzucchi SE. Use of metformin in the setting of mild-to-moderate renal insufficiency. Diabetes Care. 2011 Jun;34(6):1431-7. doi: 10.2337/dc10-2361. No abstract available. PMID 21617112
- [Background] Inzucchi SE, Lipska KJ, Mayo H, Bailey CJ, McGuire DK. Metformin in patients with type 2 diabetes and kidney disease: a systematic review. JAMA. 2014 Dec 24-31;312(24):2668-75. doi: 10.1001/jama.2014.15298. PMID 25536258
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Goldenberg R, Punthakee Z. Definition, classification and diagnosis of diabetes, prediabetes and metabolic syndrome. Can J Diabetes. 2013 Apr;37 Suppl 1:S8-11. doi: 10.1016/j.jcjd.2013.01.011. Epub 2013 Mar 26. No abstract available. PMID 24070969
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Segal RJ, Reid RD, Courneya KS, Sigal RJ, Kenny GP, Prud'Homme DG, Malone SC, Wells GA, Scott CG, Slovinec D'Angelo ME. Randomized controlled trial of resistance or aerobic exercise in men receiving radiation therapy for prostate cancer. J Clin Oncol. 2009 Jan 20;27(3):344-51. doi: 10.1200/JCO.2007.15.4963. Epub 2008 Dec 8. PMID 19064985
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Background] Antuna-Puente B, Disse E, Rabasa-Lhoret R, Laville M, Capeau J, Bastard JP. How can we measure insulin sensitivity/resistance? Diabetes Metab. 2011 Jun;37(3):179-88. doi: 10.1016/j.diabet.2011.01.002. Epub 2011 Mar 23. PMID 21435930
- [Background] Borai A, Livingstone C, Kaddam I, Ferns G. Selection of the appropriate method for the assessment of insulin resistance. BMC Med Res Methodol. 2011 Nov 23;11:158. doi: 10.1186/1471-2288-11-158. PMID 22112229
- [Background] Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ. Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans. J Clin Endocrinol Metab. 2000 Jul;85(7):2402-10. doi: 10.1210/jcem.85.7.6661. PMID 10902785
- [Background] Riediger ND, Clara I. Prevalence of metabolic syndrome in the Canadian adult population. CMAJ. 2011 Oct 18;183(15):E1127-34. doi: 10.1503/cmaj.110070. Epub 2011 Sep 12. PMID 21911558
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Derived] Roy S, Malone S, Grimes S, Morgan SC. Impact of Concomitant Medications on Biochemical Outcome in Localised Prostate Cancer Treated with Radiotherapy and Androgen Deprivation Therapy. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):181-190. doi: 10.1016/j.clon.2020.09.005. Epub 2020 Sep 29. PMID 32994091